CLINICAL TRIAL: NCT00328302
Title: Studies of Early Diabetic Glomerulopathy-the Relation Between Histopathology, Kidney Function and Metabolic Control. Natural History and Effect of ARB
Brief Title: Diabetes Type 1, Treatment Study Atacand/Placebo After Kidney Biopsy
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Karolinska University Hospital (Other)
Collaborators: AstraZeneca (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SH-AHM-0044-01
Record Dates: First submitted 2006-05-18; First posted 2006-05-19 (Estimated); Last update posted 2006-05-19 (Estimated); Status verified 2000-06

CONDITIONS: Diabetes, Type I
Keywords: Diabetes; Kidney function; 24 ambulatory blood pressure; Kidney biopsy
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Diabetes Mellitus | interventions — candesartan

INTERVENTIONS:
Drug: Candesartan
Drug: Placebo

SUMMARY:
The type 1 diabetes patients who were still normoalbuminuric and normotensive, after 17 years duration and a second research kidney biopsy, could enter the double blind treatment study of Atacand or Placebo.

The treatment study continues for five years treatment and ends with a third kidney biopsy.

The study hypothesis is that the effect of ARB during 5 years on the histopathology are more pronounced than the effect on histopathology of placebo.

DETAILED DESCRIPTION:
46 patients performed a first kidney biopsy between 1992-1994. After 6 years 29 accepted to perform a second biopsy. During the follow-up 10 patients developed complications i.e. hypertension or microalbuminuria. 7 of the patients got treatment during follow up and 3 started the treatment after the second biopsy. 19 patients with two kidney biopsies were still normoalbuminuric and normotensive. 13 of them entered the double-blind treatment study of Atacand or Placebo. 6 denied to participate in the treatment study.

The treatment study will continue for 5 years and will end with a third kidney biopsy. Also the rest of the patients that have done 2 kidney biopsies will be asked to perform a third biopsy.

ELIGIBILITY:
Inclusion Criteria:

* Diabetes type 1 patient
* Normotensive
* Normoalbuminuric
* Signed informed consent
* Female and male
* Over 17 years of age
* Diabetes duration over 10 years

Exclusion Criteria:

* Hypertension
* Microalbuminuria
* Pregnancy
* Lactation
* Reduced kidney function
* Artery stenosis
* Kidney transplantation
* Allergy to the medication in the study
* Reduced liver function
* Alcohol or drug abuse
* Participation in another drug or clinical test during last 30 days
* Severe diseases i.e. malignancy
* Previously enrolment of the present study

Ages: 17 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 13
Dates: Start 2000-09; Study Completion 2006-04

PRIMARY OUTCOMES:
Basement membrane thickness
Mesangial expansion

SECONDARY OUTCOMES:
Hypertension
Microalbuminuria
Kidney Function
24 hour ambulatory blood pressure

CONTACTS AND LOCATIONS:
Overall Officials: Nina ES Perrin, PhD-student, Principal Investigator — Karolinska University Hospital, Huddinge, B57, Childrens Hospital, 141 86 Stockholm; Ulla B Berg, Professor, Study Director — Karolinska University Hospital, B57, Childrens Hospital, 141 86 Stockholm, Sweden
Locations (1):
- Childrens Hospital, Karolinska University Hospital, Huddinge, Stockholm, Sweden

REFERENCES:
- [Derived] Perrin NE, Jaremko GA, Berg UB. The effects of candesartan on diabetes glomerulopathy: a double-blind, placebo-controlled trial. Pediatr Nephrol. 2008 Jun;23(6):947-54. doi: 10.1007/s00467-008-0745-x. PMID 18270751